CLINICAL TRIAL: NCT07024017
Title: The Acute Effects of Dynamic Stretching and Foam Rolling on Peripheral Oxygenation and Hamstring Flexibility in in Healthy Individuals With Hamstring Tightness: A Randomized Controlled Assessor Blinded Trial
Brief Title: Dynamic Stretching vs. Foam Rolling: Effects on Hamstring Flexibility and Muscle Oxygenation in Tight Hamstrings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pelin Pişirici (Other)
Responsible Party: Sponsor-Investigator, Pelin Pişirici, Assistant Professor, PT, PhD, Bahçeşehir University
Organization: Bahçeşehir University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YYLT-2025
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Hamstring Contractures; Muscle Relaxation; Muscle Tightness
Keywords: myofascial release; moxy; active knee extansion test; warm-up; Near-Infrared Spectroscopy

STUDY DESIGN:
Intervention Model Description: Participants with hamstring tightness will be randomly assigned to one of three groups: a foam rolling group, a dynamic stretching group, or a control group.
  Before the intervention, baseline assessments will include measurements of muscle oxygenation and the Active Knee Extension test to determine initial hamstring flexibility.
  After the pre-intervention evaluation, participants in the dynamic stretching group will perform a standardized series of dynamic stretching exercises, while those in the foam rolling group will apply self-administered myofascial release using a foam roller. The control group will not receive any intervention but will rest for the same duration to ensure consistency in time allocation.
  Post-intervention assessments, including measurements of muscle oxygenation and the Active Knee Extension test, will be conducted immediately after the intervention and again ten minutes later to evaluate both the immediate and short-term effects.
Who Masked: Outcomes Assessor
Masking Description: Assessor will be blind to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foam Roller (Experimental): For the foam rolling intervention, participants were positioned in an upright seated posture with the foam roller placed under the right thigh. The right leg remained extended, while the left leg was crossed over the right knee for added stability. The foam rolling movement began at the area behind the knee and progressed slowly toward the ischial tuberosity, then returned to the starting point in a continuous back-and-forth rolling pattern.
  Interventions: Device: Foam roller
- Dynamic Strecth (Experimental): The dynamic stretching protocol consisted of 10 different exercises performed over a total duration of 10 minutes at moderate to high intensity.
  Interventions: Other: dynamic stretch
- Control Group (No Intervention): The control group will not receive any intervention and will rest for the same duration.

INTERVENTIONS:
Device: Foam roller — FR will be applied to each hamstring muscle for 3 minutes per leg, totaling 6 minutes. The pressure was self-regulated by participants, who are instructed to apply as much body weight as tolerable. The rolling frequency is maintained at approximately 0.5 Hz, corresponding to one complete rolling cycle every 2 seconds. Before the intervention, participants will receive verbal and visual instructions to ensure correct execution.
  Arms: Foam Roller
Other: dynamic stretch — 10 different exercises will be performed over a 13-meter distance, with a 10-second rest period between exercises.
  During the session, participants will receive verbal feedback to ensure proper posture and technique. Exercises will be video recorded and shared with participants for review and consistency.
  Arms: Dynamic Strecth

SUMMARY:
Hamstring muscle flexibility plays a vital role in functional movement and in the prevention of injuries. Reduced flexibility of the hamstring muscles is common and can lead to biomechanical dysfunctions, a limited range of motion, and poor posture. Interventions such as stretching exercises and myofascial release techniques are widely used to improve muscle flexibility. Dynamic stretching, which involves active muscle movements, has been shown to significantly enhance flexibility and may be more effective than static stretching. The use of a foam roller, which is a self-applied myofascial release technique, also improves flexibility and may offer additional benefits by increasing fascial mobility without impairing muscle strength.

Peripheral muscle oxygenation reflects a muscle's ability to utilize oxygen and is increasingly used to assess physical performance and fatigue. Although some studies suggest that stretching exercises and foam roller applications may improve peripheral muscle oxygenation, the evidence remains limited. This study aimed to compare the effects of a single session of isolated dynamic stretching and foam roller application on hamstring muscle flexibility and muscle oxygenation. The hypothesis proposed that dynamic stretching would be more effective than foam roller application in enhancing muscle oxygenation, while both interventions would similarly improve muscle flexibility.

DETAILED DESCRIPTION:
Muscle flexibility is defined as the capacity of muscle tissue to elongate and is considered one of the key components in maintaining physical fitness. The hamstring muscles are primarily responsible for knee flexion and play a crucial role in the proper execution of functional activities. Reduced flexibility in the hamstring muscles is among the most commonly observed musculoskeletal issues, both in the general population and in athletes.

Insufficient flexibility may lead to impairments in lower extremity biomechanics, potentially resulting in various dysfunctions. A loss of hamstring flexibility limits the range of motion in the knee joint and is a critical factor that increases the risk of injury. This may occur due to passive shortening from postural adaptations or active shortening caused by muscle spasms and contractions. Decreased flexibility negatively affects posture, lower extremity mobility, and gait patterns. It may also lead to strength imbalances, overuse syndromes, and inefficient movement patterns.

Hamstring tightness can be prevented through appropriate interventions. The relative stiffness of structures such as soft tissues, joint capsules, muscles, and fascia can directly influence muscle flexibility. The myofascia surrounding the muscle is a type of connective tissue that can restrict joint range of motion and reduce muscular strength and endurance in cases of inflammation, immobilization, or tissue damage. Clinicians employ various manual techniques and stretching exercises to bring about therapeutic changes in these tissues, including osteopathic mobilizations, structural integration, massage, muscle energy techniques, and instrument-assisted soft tissue mobilizations.

Stretching exercises are among the most common interventions used to increase hamstring flexibility. When applied regularly, these exercises have been shown to enhance muscle length and elasticity. They are also fundamental components of pre-exercise warm-up routines. Dynamic stretching involves controlled movements that allow the opposing muscle to elongate throughout its full range of motion without holding a static end position, while the target muscle contracts. Studies have shown that even a single session of dynamic stretching can significantly improve hamstring flexibility. In individuals with hamstring tightness, dynamic stretching has been found to be more effective than static stretching.

As an alternative, self-administered myofascial release techniques are also widely used. These techniques are most commonly performed using foam rollers and work similarly to traditional manual myofascial release methods. The pressure is applied with the help of body weight, providing direct and continuous compression to the soft tissue. This pressure enhances fascial mobility, increases joint range of motion, raises fascial temperature through friction, and reduces extracellular matrix viscosity. These changes help to resolve adhesions between fascial layers and restore tissue extensibility. Foam roller applications have been shown to acutely improve hamstring flexibility without negatively affecting muscle strength and may be more effective than both static stretching and dynamic stretching exercises.

Peripheral muscle oxygenation refers to the level of oxygenation in muscles distant from central circulation and reflects the muscle's oxygen uptake and utilization capacity. Measuring oxygen saturation in the hamstring muscles provides direct insight into their metabolic performance. Recently, such measurements have become increasingly used to analyze training load, fatigue, and injury risk. However, findings on the effects of stretching or myofascial release on peripheral muscle oxygenation remain limited. It has been suggested that both static stretching and dynamic stretching during warm-ups may increase intramuscular oxygen availability. Some studies have shown that oxygen saturation levels are higher after dynamic stretching compared to static stretching. Furthermore, combining stretching with foam roller applications has been shown to further increase muscle oxygenation, suggesting that the oxygen supplied exceeds the intramuscular oxygen demand. Nevertheless, there is a need for studies that investigate the isolated effects of dynamic stretching and foam roller application.

The aim of this study was to compare the effects of a single, isolated session of dynamic stretching and foam roller application on hamstring flexibility and peripheral muscle oxygenation. The hypothesis was that, in healthy individuals with hamstring tightness, dynamic stretching would be more effective than foam roller application in increasing muscle oxygenation, while both interventions would have similar effects on flexibility.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged between 18 and 35 years
* Both male and female participants
* Absence of any known health conditions
* Hamstring tightness defined as ≥20° of knee flexion angle in Active Knee Extension test

Exclusion Criteria:

* Any neuromuscular or orthopedic disorders affecting the lower extremities
* Circulatory or vascular problems
* Respiratory or cardiovascular diseases
* Renal failure
* Presence of pain during measurements or exercise protocols
* Excessive skin sensitivity or active skin infection
* History of intense physical activity within the last 48 hours

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Muscle Oxygenation Assessment | baseline, immediately after the intervention, ten minutes after the baseline
  Muscle oxygenation will be assessed using the MOXY Monitor, which is a portable, wireless device based on near-infrared spectroscopy. The monitor will be placed on the belly of the right biceps femoris muscle and secured with an opaque elastic band to prevent interference from ambient light.
  Measurements will be taken five minutes before and five minutes after the intervention session. During each measurement period, the device will record data for sixty seconds, and the average muscle oxygen saturation value over this period will be used for analysis.

SECONDARY OUTCOMES:
Active Knee Extension (AKE) Test | baseline, immediately after the intervention, ten minutes after the baseline
  The Active Knee Extension test will be used as a secondary outcome measure to assess hamstring muscle flexibility. Participants will lie in a supine position with the leg that is not being tested fully extended. The leg being tested will be positioned in ninety degrees of hip flexion using a wooden box to stabilize the pelvis and the thigh.
  Participants will actively extend the knee until a visible muscle spasm or twitch occurs. They will then slowly lower the leg until the movement stops. At that point, the knee flexion angle will be measured using a goniometer. The average value from three trials will be recorded for each leg.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Akgöl, PT, Principal Investigator — Bahcesehir University, Graduate Education Institute, Physiotherapy and Rehabilitation, Master of Science Program; Pelin Pişirici, PT, PhD, Study Director — Bahcesehir University, Faculty of Health Sciences
Locations (1):
- Bahcesehir University, Istanbul, Beşiktaş, Turkey (Türkiye)